CLINICAL TRIAL: NCT03430505
Title: Effects of Noninvasive Ventilation Compared to Salbutamol in Respiratory Mechanics and Lung Function of Asthmatics After Bronchoprovocation: Randomized Cross-over Trial
Brief Title: Effects of Noninvasive Ventilation Compared to Salbutamol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Evelim Leal de Freitas Dantas Gomes, PT, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OEP Asthma
Record Dates: First submitted 2018-01-31; First posted 2018-02-13 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: Asthma, noninvasive ventilation
MeSH Terms: conditions — Asthma | interventions — Continuous Positive Airway Pressure; Albuterol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilevel (Active Comparator): Bilevel 10 minutes after bronchoprovocation with saline solution 4.5%. IPAP 12 and EPAP 8
  Interventions: Device: Bilevel
- Albuterol (Active Comparator): 400micrograms after bronchoprovocation with saline solution 4.5%.
  Interventions: Drug: Albuterol

INTERVENTIONS:
Device: Bilevel — Basal respiratory mechanics in spontaneous breathing will be analyzed by optoeletronic plethismography (OEP), followed by bronchial provocation with hypertonic saline solution 4.5%, another 45-second OEP uptake, IPAP 12 and EPAP 8 bilevel applied for 10 minutes, and a new uptake. All abstractions are preceded by a forced and slow spirometry maneuver. The entire procedure takes 1 hour.
  Arms: Bilevel
Drug: Albuterol — Basal respiratory mechanics in spontaneous breathing will be analyzed by optoeletronic plethismography (OEP), followed by bronchial provocation with hypertonic saline solution 4.5%, another 45-second OEP uptake, 400 micrograms inhaled Albuterol, and a new uptake. All abstractions are preceded by a forced and slow spirometry maneuver. The entire procedure takes 1 hour.
  Arms: Albuterol

SUMMARY:
Asthma is a chronic inflammatory disease characterized by recurrent and reversible episodes of airway obstruction. Drug treatment usually includes inhaled corticosteroids and bronchial dilators, which often do not have adequate adherence. These acute episodes of bronchoconstriction can most often occur with hyperinflation and for decades the mechanisms that lead to hyperinflation have been studied, as well as increasingly modern ways of evaluating and treating these mechanisms. Noninvasive ventilation is increasingly occupying its space as a non-pharmacological resource in the treatment of asthma, initially as an adjunct in an attempt to help medication have its effect reached in the crisis, but this feature has been showing signs of having an even greater action which can even collaborate in reversing the crisis by not only giving time for pharmacological action. Recognizing these potential effects of this widely used resource and understanding its action on lung function and the reversal of exacerbation is part of this scientific process.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease characterized by recurrent episodes of reversible airway obstruction. The drug treatment typically includes inhaled steroids and bronco dilators. These acute episodes of bronchoconstriction can, for the most part, attend with hyperinflation, the hyperinflation and the consequent increase of functional residual capacity (FRC) inspiratory muscle activation in phase before the expiratory lung elastic equilibrium and rib cage.

Some studies reports the injury to respiratory function that causes acute hyperinflation with a reduction of the contribution of the abdominal compartment and increased assistance from the chest compartment, thereby reducing the efficiency mechanics of the diaphragm in response to decreased your stamping area. As a result of this disadvantage and mechanics "reduction of curvature" of the diaphragm expiratory muscle activation occurs in an attempt to restore the original mechanics and thus your primary function.

Some studies have investigated the effects of bronchoconstriction in recruitment of the respiratory muscles and respiratory mechanics of patients susceptible to asthma. As asthma has distinct characteristics in crisis and in stable phase, testing of bronchial provocation test have been part of the studies allowing assessment in different physiological conditions, close to an acute condition without necessarily a crisis and insufficiency that would make it really an assessment respiratory kinematics and the involvement of the thoracic and abdominal compartments in each of these phases and mainly in front of any therapy.

Bronchial provocation tests are safe once they cause the release of endogenous mediators that cause the bronchial smooth muscle contraction causing narrowing of the airway, but as your sensitivity is reduced your action is completely reversed with use of bronchodilator and the positive response to these tests that can be performed by exercise or inhaling hypertonic solution 4.5% reflect a inflammation of the Airways.

The interest in the implementation of non-pharmacological therapies and especially the knowledge of resources used often to relieve the overload of respiratory muscles in patients with obstructive, since the Decade of 80, has been demonstrating that the use of expiratory positive pressure can reduce muscle work and reduce the volume of expiratory reserve contributing to deflation.

Most recently the bronchodilator effect of CPAP mediated by autonomic receptors stretch lung. What we need to know is the effect of non-invasive ventilation with two levels of pressure can in addition to trigger this neural reflex, can still promote a kinematics similar to produced by bronchodilator seen through optoelectronics plethysmography (OEP).

The Optoelectronics Plethysmography (OEP) has made possible the exploitation of Thoracoabdominal movement by magazines, reporting especially changes in total volume of the chest wall during any intervention as the NIV.

The OEP is an innovative method of indirect measurement of pulmonary ventilation, and your application can be used in different health conditions, like asthma and neuromuscular diseases, with different protocols. Is a non-invasive method and measurement of non-ionizing lung volumes, able to detect small movements of the chest wall during breathing through the analysis of reflective markers attached to the chest wall of the individual; There is no need to use mouthpiece, nasal clip or other connector of the equipment to the individual; the calibration is fast and without the participation of the subject.

Since the NIV with bi-level pressure promotes a level of inspiratory pressure that increases the expiratory ventilation and a stretch of lung receptors stimulates and bronchodilator effect, the hypothesis of this study is that the thoracic and abdominal configuration and improvement of pulmonary function after test of bronchial provocation test is considerable with the NIV compared to bronchodilator. There are no studies in the literature that discuss this subject under this optics of assessment.

The aim of this study is to evaluate the effects of the NIV in reversal of bronchial provocation test and your potential bronchodilator effect compared to the gold standard bronchodilator drug seen by thoracic and abdominal and lung function configuration.

2. General Purpose

To evaluate the responses of the thoracoabdominal configuration and the participation of the thoracic and abdominal compartments in asthmatic patients before the bronchoprovocation test and in response to pharmacological and non-pharmacological therapy.

2.1. Specific objectives

* To evaluate the abdominal thoracic configuration of adolescents and young adults with stable asthma before and after bronchoprovocation
* To evaluate the effect of bronchodilator and NIV in the thoraco-abdominal configuration

  3. Materials and Methods

3.1. Kind of study

This is a randomized, crossover clinical trial in which it will be performed in two visits and evaluated the abdominal thoracic configuration before and after bronchoprovocation and after bronchodilator and non-invasive ventilation (NIV) with two levels of pressure in adolescents and young adults with asthma.

3.2. Ethical aspects

This study will be developed respecting the research standards involving human beings (Resolution CNS 466/2012) of the National Health Council, was approved by the Research Ethics Committee of the University Nove de Julho (2.130.007 / 2017). You will have your registration done at clincaltrial.gov.

3.3. Place of study and sample

The study will be developed in the Multidisciplinary Laboratory of Movement, Optical Electronic Plethysmography (OEP) and in the Functional Respiratory Evaluation Laboratory located at the Latin American Memorial Campus of the University of Nove de Julho (UNINOVE), at Francisco Matarazzo Avenue, 376, Barra Funda , Sao Paulo-SP.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 12 to 29 years
* Both sexes
* Diagnosis of asthma according to GINA
* Without deterioration in the last 30 days
* No history of respiratory infection in the last 2 months
* Comply with consent form

EXCLUSION CRITERIA:

* Use bronchodilator under 12 hours
* No understanding of the tests
* Heart condition
* Intolerance the proposed activities
* Don't have bronchodilator prescribed by doctor

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
FEV1 | Change from baseline FEV1 at 1 hour
  Spirometry
Expiratory time | Change from baseline expiratory time at 1 hour
  Optoeletronic Plethismography
Inspiratory Capacity | Change from baseline IC at 1 hour
  Spirometry

SECONDARY OUTCOMES:
Minute Volume | Change from baseline minute volume at 1 hour
  Optoeletronic Plethismography

CONTACTS AND LOCATIONS:
Overall Officials: Dirceu Costa, Doctor, Study Chair — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No